CLINICAL TRIAL: NCT00520364
Title: In Vitro Fertilization and Pregnancy After Use of Chemotherapy
Status: Terminated | Type: Observational
Why Stopped: PI left the Institution.
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, kutluk oktay, PI, New York Medical College
Other Study IDs: 0502007757
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Anti-Mullerian Hormone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- History of chemotherapy: IVF after chemotherapy
  Interventions: Other: Observation of IVF outcomes in relation to chemo history and AMH
- IVF without history of chemotherapy: IVF without history of prior chemotherapy
  Interventions: Other: Observation of IVF outcomes in relation to chemo history and AMH

INTERVENTIONS:
Other: Observation of IVF outcomes in relation to chemo history and AMH — Women undergoing IVF with or without history of chemotherapy, AMH levels compared

SUMMARY:
Objective: Chemotherapy regimens containing alkylating agents result in primordial follicle death and premature ovarian failure. Depending on the age and the type/dose of chemotherapy, some women may continue to menstruate. Our aim was to ascertain the impact of chemotherapy on ovarian reserve in patients who previously received chemotherapy by response to controlled ovarian hyper stimulation (COH) and anti-mullerian hormone (AMH) levels. Design: Prospective study with retrospective controls Materials and Methods: 45 cancer patients underwent controlled ovarian stimulation for IVF before (30 patients, 30 IVF cycles) or after (15 patients, 30 IVF cycles) chemotherapy. Patients with basal serum FSH >13mIU/mL or E2>70pg/ml were excluded. AMH was measured on previously stored serum samples from the day of initiation of the ovarian stimulation. Results: Mean ages and baseline FSH levels of pre- and postchemotherapy IVF patients were similar (36.8±0.91 vs. 36.3±1). The mean interval from completion of chemotherapy to IVF was 8.03±1.32 years (range 1-23). Of the 30 IVF cycles in post-chemotherapy patients, 22 received alkylating agents and 8 did not.

There were no significant differences between the study and control cycles regarding day-2 estradiol (E2), length of stimulation, total gonadotropin dose, and E2 on hCG day (table 2). Cycle cancellation rate was 20% and 26.67% for pre and post-chemotherapy patients, respectively. The number of oocytes retrieved and fertilized were significantly higher in pre-chemotherapy group (p<0.0001). Two clinical pregnancies were achieved in the postchemotherapy group, one ending in spontaneous abortion and the other in the delivery of a healthy baby (6.67% clinical pregnancy rate and 3.33% delivery rate per attempted cycle). All fertilized oocytes in the control group were cryopreserved at 2-pronuclei stage.

Baseline AMH levels were significantly lower in post chemotherapy IVF patients compared to those who underwent IVF prior to chemotherapy (0.270 ±0.077 vs. 0.84±0.27 ng/ml, p=0.03). In the pre-chemotherapy group there was a positive correlation between the AMH levels and the number of oocytes retrieved (r=0.663, p=0.004 ). This correlation was not detected in the post chemotherapy group (r=0.205).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* Histologically confirmed cancer diagnosis
* Received chemotherapy more than one year ago
* Have both ovaries
* Regular menstrual cycle
* Normal basal FSH, LH and estradiol

Exclusion Criteria:

* >42 years
* Radiation below the diaphragm
* Ovarian failure

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Response to controlled ovarian stimulation | during IVF stimulation
AMH levels | during IVF

SECONDARY OUTCOMES:
Ongoing pregnancy | after IVF

CONTACTS AND LOCATIONS:
Overall Officials: Kutluk Oktay, MD, Principal Investigator — New York Medical College
Locations (1):
- IFP, New York, New York, United States